CLINICAL TRIAL: NCT02642562
Title: Effectiveness of Intravenous Iron Treatment vs Standard Care in Patients With Heart Failure and Iron Deficiency: a Randomised, Open-label Multicentre Trial (IRONMAN)
Brief Title: Intravenous Iron Treatment in Patients With Heart Failure and Iron Deficiency: IRONMAN
Acronym: IRONMAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); Pharmacosmos A/S (Industry); British Heart Foundation (Other)
Responsible Party: Principal Investigator, Paul Kalra, Chief Investigator, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN15CA190
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Chronic Heart Failure; Iron Deficiency; Left Ventricular Systolic Dysfunction
Keywords: Intravenous iron; PROBE design
MeSH Terms: conditions — Iron Deficiencies; Ventricular Dysfunction, Left | interventions — ferric derisomaltose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (No Intervention): Participants in this arm will receive their usual care
- Standard care plus IV iron infusion (Experimental): Iron to be administered as iron (III) isomaltoside 1000 / ferric derisomaltose.
  Infused over a minimum of 15 mins for doses up to and including 1000mg, and a minimum of 30 mins for doses >1000mg
  Where Hb ≥10 g/dL, dosage according to body weight is as follows:
  Body weight <50 kg: 20 mg/kg; Body weight 50 to <70 kg: 1000 mg; Body weight ≥70 kg: 20 mg/kg up to a maximum of 1500 mg.
  Where Hb <10 g/dL, dosage according to body weight is as follows:
  Body weight <50 kg: 20 mg/kg; Body weight 50 to <70 kg: 20 mg/kg; Body weight ≥70 kg: 20 mg/kg up to a maximum of 2000 mg.
  Interventions: Drug: Ferric Derisomaltose

INTERVENTIONS:
Drug: Ferric Derisomaltose
  Other Names: Monofer
  Arms: Standard care plus IV iron infusion

SUMMARY:
This study will address whether the additional use of Intravenous (IV) iron on top of standard care will improve the outlook for patients with heart failure and iron deficiency. One group of participants will receive treatment with iron injections and the other group will not receive any iron injections.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) is a very common medical problem. Despite improvements in treatment, many patients suffer limiting symptoms of shortness of breath and fatigue. Hospitalisation for CHF is common and life expectancy reduced. Many patients with CHF have a deficiency of iron (low iron levels or cannot use iron properly), and this is associated with poorer outcomes. Some small research studies have suggested that giving patients intravenous iron improves symptoms in the short term. It is unknown, however, whether correcting iron deficiency is beneficial to patients with CHF in the long term and whether it improves life expectancy and keeps them out of hospital. This study will help us answer these key questions.

This study will address whether the additional use of Intravenous (IV) iron on top of standard care will improve the outlook for patients with heart failure and iron deficiency. One group of participants will receive treatment with iron injections and the other group will not receive any iron injections.

The study will take place in about 70 secondary care sites (hospitals) across the UK. Participants will be recruited over a period of about five years and will be followed up for a minimum of three months (average duration of about four years per participant). After the initial visits, participants will be seen every four months.

ELIGIBILITY:
Inclusion criteria

1. Age ≥18 years
2. LVEF ≤45% within the prior two years using any conventional imaging modality (this should be the most recent assessment of LVEF)
3. New York Heart Association (NYHA) class II - IV
4. Iron deficient - defined as TSAT <20% and/or ferritin <100 ug/L
5. Evidence of being in a higher risk HF group: (a) Current (with the expectation that patient will survive to discharge) or recent (within 6 months) hospitalisation for HF, OR (b) Out-patients with NT-proBNP >250 ng/L in sinus rhythm or >1,000 ng/L in atrial fibrillation (or BNP of > 75 pg/mL or 300 pg/mL, respectively)
6. Able and willing to provide informed consent

Exclusion criteria

1. Haematological criteria: ferritin >400ug/L; haemoglobin <9.0, or >13 g/dL in women or >14g/dL in men; (B12 or folate deficiency should be corrected but do not exclude the patient)
2. MDRD/CKD-EPI estimated glomerular filtration rate (eGFR) <15ml/min/1.73m2
3. Already planned to receive IV iron
4. Likely to need or already receiving erythropoiesis stimulating agents (ESA)
5. Any of the following apply: (a) planned cardiac surgery or revascularisation; (b) within 3 months of any of the following: a primary diagnosis of type 1 myocardial infarction (excluding small troponin elevations in the context of heart failure admissions), cerebrovascular accident (CVA), major CV surgery or percutaneous coronary intervention (PCI), or blood transfusion; (c) on active cardiac transplant list; (d) left ventricular assist device implanted.
6. Any of the following comorbidities: active infection (if the patient is suffering from a significant ongoing infection as judged by the investigator recruitment should be postponed until the infection has passed or is controlled by antibiotics), other disease with life expectancy of <2 years, active clinically relevant bleeding in the investigator's opinion, known or suspected gastro-intestinal malignancy
7. Pregnancy, women of childbearing potential (i.e. continuing menstrual cycle) not using effective contraception (see Appendix 3) or breast-feeding women
8. Contra-indication to IV iron in the investigator's opinion according to current approved Summary of Product Characteristics: hypersensitivity to the active substance, to Monofer® or any of its excipients (water for injections, sodium hydroxide (for pH adjustment), hydrochloric acid (for pH adjustment)); known serious hypersensitivity to other parenteral iron products; non-iron deficiency anaemia (e.g. haemolytic anaemia); iron overload or disturbances in utilisation of iron (e.g. haemochromatosis, haemosiderosis); decompensated liver disease.
9. Participation in another intervention study involving a drug or device within the past 90 days (co-enrolment in observational studies is permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1160 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
CV mortality or hospitalisation for worsening heart failure (analysis will include first and recurrent hospitalisations) | Minimum of 3 months follow-up from last patient recruited

SECONDARY OUTCOMES:
Hospitalisation for worsening heart failure (recurrent events) | Minimum of 3 months follow-up from last patient recruited
CV hospitalisation (first event) | Minimum of 3 months follow-up from last patient recruited
CV death or hospitalisation for heart failure analysed as time to first event | Minimum of 3 months follow-up from last patient recruited
Overall Score from Minnesota Living with Heart Failure | At 4 months
Cardiovascular mortality | Minimum of 3 months follow-up from last patient recruited
Overall EQ-5D VAS | At 4 months
Overall EQ-5D index | At 4 months
CV mortality or hospitalisation for major CV event (stroke, MI, heart failure) (first event) | Minimum of 3 months follow-up from last patient recruited
All-cause mortality | Minimum of 3 months follow-up from last patient recruited
All-cause hospitalisation (first event) | Minimum of 3 months follow-up from last patient recruited
Combined all-cause mortality or first all-cause unplanned hospitalisation | Minimum of 3 months follow-up from last patient recruited
Physical domain of QoL (Minnesota Living With Heart Failure) | At 4 months
Physical domain of QoL (Minnesota Living With Heart Failure) | At 20 months
Overall EQ-5D VAS | At 20 months
Overall EQ-5D index | At 20 months
Overall Score from Minnesota Living With Heart Failure | At 20 months
Days dead or hospitalised | At 36 months
Quality-adjusted days alive and out of hospital | At 12 months
6 minute walk test | At 4 months
6 minute walk test | At 20 months
Death due to infection | Minimum of 3 months follow-up from last patient recruited
Hospitalisation primarily for infection (first event) | Minimum of 3 months follow-up from last patient recruited

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Boon, Study Chair — Chair of Steering Committee (Retired)
Locations (72):
- United Kingdom (72):
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospital Monklands, Airdrie
  - Antrim Area Hospital, Antrim
  - Wansbeck General Hospital, Ashington
  - Barnet Hospital, Barnet
  - Basildon University Hospital, Basildon
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Royal Victoria Hospital, Belfast
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - Princess of Wales Hospital, Bridgend
  - Royal Sussex County Hospital, Brighton
  - Bristol Royal Infirmary, Bristol
  - Broomfield Hospital, Chelmsford
  - Chesterfield Royal Hospital, Chesterfield
  - St. Richard's Hospital, Chichester
  - University Hospital Coventry, Coventry
  - Croydon University Hospital, Croydon
  - Darlington Memorial Hospital, Darlington
  - Doncaster Royal Infirmary, Doncaster
  - Ninewells Hospital, Dundee
  - Ulster Hospital, Dundonald
  - Eastbourne District General Hospital, Eastbourne
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Glasgow Royal Infirmary, Glasgow
  - Golden Jubilee National Hospital, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Harefield Hospital, Harefield
  - Wycombe General Hospital, High Wycombe
  - Castle Hill Hospital, Hull
  - Raigmore Hospital, Inverness
  - West Middlesex University Hospital, Isleworth
  - University Hospital Crosshouse, Kilmarnock
  - Kingston Hospital, Kingston upon Thames
  - Victoria Hospital, Kirkcaldy
  - Forth Valley Royal Hospital, Larbert
  - Glenfield Hospital, Leicester
  - Aintree University Hospital, Liverpool
  - Liverpool Heart and Chest Hospital, Liverpool
  - University Hospital Llandough, Llandough
  - Royal Glamorgan Hospital, Llantrisant
  - Guy's and St. Thomas' Hospital, London
  - Hammersmith Hospital (Imperial College), London
  - King's College Hospital, London
  - North Middlesex University Hospital, London
  - St. Bartholomew's Hospital, London
  - University College London Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Wythenshawe Hospital, Manchester
  - Royal Gwent Hospital, Newport
  - Nottingham University Hospital, Nottingham
  - Royal Oldham Hospital, Oldham
  - John Radcliffe Hospital, Oxford
  - Royal Alexandra Hospital, Paisley
  - Poole Hospital, Poole
  - Queen Alexandra Hospital, Portsmouth
  - Salford Royal Hospital, Salford
  - Salisbury District Hospital, Salisbury
  - Northern General Hospital, Sheffield
  - University Hospital Southampton, Southampton
  - Southend University Hospital, Southend
  - Royal Stoke University Hospital, Stoke-on-Trent
  - City Hospitals Sunderland, Sunderland
  - Morriston Hospital, Swansea
  - Great Western Hospital, Swindon
  - St. George's Hospital, Tooting
  - Torbay Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Watford General Hospital, Watford
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Applications for data access will be considered when analysis of the main pre-specified endpoints, sub-groups and sub-studies, and other sub-analyses have been completed.
Supporting Information: Study Protocol, SAP
Time Frame: Applications for access will be considered when analysis of the main pre-specified endpoints, sub-groups and sub-studies, and other sub-analyses have been completed.
Access Criteria: Applications for access will be reviewed by the study Steering Committee.

REFERENCES:
- [Derived] Sze S, Squire I, Kalra PR, Cleland JG, Petrie MC, Kalra PA, Ahmed F, Banerjee P, Boos CJ, Chapman C, Cowburn PJ, Dixon L, Duckett S, Lane R, Foley P, Lang NN, Lyons K, Ray R, Schiff R, Thomson EA, Robertson M, Ford I; IRONMAN Study group. Age-stratified effects of intravenous ferric derisomaltose in heart failure with iron deficiency: insights from the IRONMAN trial. Heart. 2025 Jun 13;111(13):634-641. doi: 10.1136/heartjnl-2024-324908. PMID 39938943
- [Derived] Foley PW, Kalra PR, Cleland JGF, Petrie MC, Kalra PA, Squire I, Campbell P, Chapman C, Donnelly P, Graham F, Hannah A, Lang NN, Matthews I, Leslie SJ, Pellicori P, Piper S, Ray R, Savage HO, Spencer C, Walsh J, Wong YK, Ford I; on behalf of the IRONMAN Study Group. Effect of correcting iron deficiency on the risk of serious infection in heart failure: Insights from the IRONMAN trial. Eur J Heart Fail. 2025 Jan;27(1):166-173. doi: 10.1002/ejhf.3504. Epub 2024 Oct 25. PMID 39453738
- [Derived] Cleland JGF, Pellicori P, Graham FJ, Lane R, Petrie MC, Ahmed F, Squire IB, Ludman A, Japp A, Al-Mohammad A, Clark AL, Szwejkowski B, Critoph C, Chong V, Schiff R, Nageh T, Glover J, McMurray JJV, Thomson EA, Robertson M, Ford I, Kalra PA, Kalra PR; IRONMAN Study Group. Adjudication of Hospitalizations and Deaths in the IRONMAN Trial of Intravenous Iron for Heart Failure. J Am Coll Cardiol. 2024 Oct 29;84(18):1704-1717. doi: 10.1016/j.jacc.2024.08.052. PMID 39443013
- [Derived] Kalra PR, Cleland JGF, Petrie MC, Thomson EA, Kalra PA, Squire IB, Ahmed FZ, Al-Mohammad A, Cowburn PJ, Foley PWX, Graham FJ, Japp AG, Lane RE, Lang NN, Ludman AJ, Macdougall IC, Pellicori P, Ray R, Robertson M, Seed A, Ford I; IRONMAN Study Group. Intravenous ferric derisomaltose in patients with heart failure and iron deficiency in the UK (IRONMAN): an investigator-initiated, prospective, randomised, open-label, blinded-endpoint trial. Lancet. 2022 Dec 17;400(10369):2199-2209. doi: 10.1016/S0140-6736(22)02083-9. Epub 2022 Nov 5. PMID 36347265
- [Derived] Kalra PR, Cleland JG, Petrie MC, Ahmed FZ, Foley PW, Kalra PA, Lang NN, Lane RE, Macdougall IC, Pellicori P, Pope MTB, Robertson M, Squire IB, Thomson EA, Ford I. Rationale and design of a randomised trial of intravenous iron in patients with heart failure. Heart. 2022 Nov 24;108(24):1979-1985. doi: 10.1136/heartjnl-2022-321304. PMID 35948408